CLINICAL TRIAL: NCT01264809
Title: Does Exercise Consultation Have a Realistic Chance of Increasing the Physical Activity Level of Type 2 Diabetes Patients in Real Life?
Brief Title: Exercise Consultation for Type 2 Diabetes Patients in Real Life
Acronym: APDT 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: Clinique Antilles-Guyane (Other)
Responsible Party: FAGOUR Cédric, CHU de Fort-de-France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 09/B/07; 2010-A00450-39 (Other: Afssaps- French Health Products Safety Agency)
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A : immediate physical activity counseling (Experimental): Participants randomized in the experimental group (group A) will receive physical activity counseling during a one-to-one consultation at both baseline and 3 months.
  Interventions: Behavioral: Specific consultation for physical activity counseling
- B : later physical activity counseling (Active Comparator): Exercise consultation will be realised only at 3 months in the control group(group B). Furthermore, patients of group B will not received any physical activity counseling at baseline.
  Interventions: Behavioral: Consultation for physical activity counseling

INTERVENTIONS:
Behavioral: Specific consultation for physical activity counseling — Specific consultation
  Arms: A : immediate physical activity counseling
Behavioral: Consultation for physical activity counseling — Specific consultation
  Arms: B : later physical activity counseling

SUMMARY:
The prevalence of type 2 diabetes is high and expected to increase dramatically in worldwide, in France and especially in the French West Indies.This chronic disease is associated with premature mortality and various debilitating complications which can be prevented by optimal control of glycaemia, blood pressure and lipids. Diabetes management includes lifestyle modification and medication. Despite numerous studies supporting the benefits of frequent physical activity for people with Type 2 diabetes, an estimated 60±80% of this population remain sedentary. Promotion of physical activity in current diabetes care seems to be inadequate.

The aim of this randomized controlled trial is to evaluate the medium-term effectiveness (after 3 and 6months) of exercise consultation in promoting physical activity in outpatients with Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 DM diagnosed within 10 years prior the inclusion
* 18-70 years old
* Signed written informed consent
* Diabetes treatment regimens :

  * diet only
  * oral antidiabetic drug
  * oral antidiabetic drugs with long acting insulin analog
  * oral antidiabetic drugs with GLP 1 analog

Exclusion Criteria:

* Minors
* Patients with concurrent medical conditions preventing exercise
* Pregnancy or intention to become pregnant during the study
* Inability to read and write French
* History of participating in our education program during the past two years
* Usual sporty activities
* Change in diabetes treatment during the three months prior to study enrollment
* No written informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Change in daily physical activity measured by SenseWear Pro3 Armband®. Participants were instructed to wear the monitor for seven days during all waking hours except bathing. | 3 months

SECONDARY OUTCOMES:
Benefits obtained after the physical activity counseling | 6 months
  The secondary outcome of this study is to compare the benefits obtained 3 and 6 mounths after the physical activity counseling on :
  * Quality of life scores
  * Anthropometric measurement and Body Mass Index (BMI)
  * Body composition measurement
  * Hand grip strength
  * Blood pressure
  * Glycaemic control and cholesterol
  * Medication

CONTACTS AND LOCATIONS:
Overall Officials: Cédric FAGOUR, MD, Principal Investigator — CHU de Fort-de-France
Locations (2):
- France (2):
  - CHU de Fort-de-France- Hôpital Pierre Zobda Quitman, Fort-de-France, Martinique
  - CHU de Bordeaux - Hôpital Haut Lévêque, Pessac